CLINICAL TRIAL: NCT01498055
Title: A Randomized Controlled Trail on the Efficacy and Safety of Autologous Cytokine-induced Killer (CIK) Cells Infusion Treatment in Advanced Primary Lung Cancer
Brief Title: Autologous CIK Cells Infusion for the Treatment of Lung Cancer: a Randomized Controlled Study
Acronym: CIK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Gong Liang, MD, Third Military Medical University
Other Study IDs: GLiang
Record Dates: First submitted 2011-11-24; First posted 2011-12-23 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2011-12

CONDITIONS: Lung Cancer
Keywords: lung cancer; CIK cells; therapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The one-time folic acid sodium anticoagulation vacuum picks bag, through the venous blood sampling 60 ml. When blood alcohol on parts of the need blood disinfects processing. After the department shows will seal in a sterile bag, 16-21 degrees Celsius save, and transported to a cell biological treatment as soon as possible a follow-up operation center GMP laboratory.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CIK therapy group
- control group

SUMMARY:
To study the efficacy and safety of autologous CIK cells infusion for the treatment of lung cancer.

DETAILED DESCRIPTION:
A randomized controlled trail on the efficacy and safety of autologous cytokine-induced killer (CIK) cells infusion treatment in advanced primary lung cancer

ELIGIBILITY:
Inclusion Criteria:

* 18~70 year old, KPS score >50 points, estimate survival > 3 months;
* Primary lung cancer patients after chemotherapy or radiation therapy;
* Primary lung cancer patients after targeted therapy;
* Primary lung cancer patients with lung function can not accept operation or unwilling to operation;
* Primary lung cancer recurrence or surgery can't complete resection;
* Primary lung cancer patients after intervention therapy(I125 implanted, freezing, rf, etc.);
* No serious mental illness and no serious heart, liver, kidney diseases, unincorporated other potentially lethal diseases;
* Patients Voluntary attempt, and informed consent.

Exclusion Criteria:

* History of cardiovascular disease: congestive heart failure > New York heart association (NYHA) level II, unstable angina patients (resting when the angina symptoms) or new happen angina pectoris (recent 3 months) or recent 6 months of myocardial infarction;
* Cachexia; or other deadly diseases;
* Liver function laboratory ALT, AST more than normal limits on 2.0 times ; Or kidney TBIL, BUN more than normal limits on 1.0 times , or Cr more than normal upper limit;
* Active infection;
* Pregnant or lactating women
* At present Is receiving other cancer treatment (such as chemotherapy, radiation therapy, chemotherapy, immunosuppressants and thrombosis, targeted agents);
* Now or recently will join another experimental clinical study ;
* Other situations that the researchers considered unsuitable for this study (such as mental illness, drug abuse, HIV infections, etc.), or influence on the results of clinical trials for analysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary lung cancer diagnosis (including small cell lung cancer, lung adenocarcinoma, lung squamous cell carcinoma and large cell carcinoma) patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rates (DCR) | From 12-2011 to 12-2013
  Lung lesions of disease control rates DCR (CR + PR + SD), according to solid tumor response evaluation standard (response evaluation criteria in solid tumors, RECIST) standard

SECONDARY OUTCOMES:
Overall Survival(OS) | 2 years
  Disease progression-free surial (Progression-Free Srvival, PFS) with observations

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Zhou, Study Chair — Southwest Hospital Third Military University
Locations (1):
- Liang Gong, Chongqing, Chong Qing, China